CLINICAL TRIAL: NCT01517048
Title: Brain-Derived Neurotrophic Factor in Obesity and Neurocognitive Function
Brief Title: Brain-Derived Neurotrophic Factor in Obesity and Brain Function
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120051; 12-CH-0051
Record Dates: First submitted 2012-01-24; First posted 2012-01-25 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-12-12

CONDITIONS: Obesity; Genetic Disorder; Mental Retardation; Developmental Delay
Keywords: Body Composition; Obesity; Overweight; Energy Homeostasis; Nociception; Prader-Willi Syndrome; Genetic Disorder; Healthy Volunteer; HV
MeSH Terms: conditions — Obesity; Genetic Diseases, Inborn; Intellectual Disability; Learning Disabilities; Overweight; Prader-Willi Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

SUMMARY:
Background:

- Prader-Willi syndrome (PWS) and MC4R genetic mutations are two conditions that can cause problems with appetite regulation. People with PWS often have behavior and thinking problems. People with MC4R mutations may have problems with attention. These problems may be related to Brain-Derived Neurotrophic Factor (BDNF), a protein that is important for brain development. Researchers want to study people with PWS and MC4R mutations to see how BDNF is involved in these conditions. Specifically, body weight and brain function will be studied, and compared with healthy volunteers.

Objectives:

- To study how BDNF affects body weight and brain function in people with PWS and MC4R mutations.

Eligibility:

* Individuals of any age who have Prader-Willi syndrome or MC4R genetic mutations.
* Healthy volunteers of any age to act as control participants.

Design:

* Participants will be screened with a medical history and physical exam. Height, weight, and waist/hip circumferences will be measured. Blood samples will be taken for genetic and other tests.
* Participants will fill out questionnaires about eating habits, pain perception, and sleep behavior.
* Participants will keep a 3-day food diary to record all food and drinks eaten.
* Tests and questionnaires will be given to study thinking, speech, movement, behavior, and mood. Some tests will be done on a computer; other tests will be on paper. Tests may also involve performing tasks with blocks and other objects.
* Participants may have other tests as directed. These will include hot and cold sensitivity tests, imaging studies like x-rays, and measurements of body fat and water content.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
Brain-derived neurotrophic factor (BDNF) is a protein that is important in nervous system development and function. BDNF also appears to function downstream of the leptin-melanocortin signaling pathway to control appetite. In both animals and humans, diminished BDNF function is associated with hyperphagia, obesity, and neurocognitive deficits. We propose to study BDNF in two hyperphagic disorders: Prader-Willi syndrome and MC4R function-altering mutations. We hypothesize that patients with PWS may have increased BDNF during infancy, followed by a decline in BDNF that precedes the onset of hyperphagia and persists after the onset of obesity. We hypothesize that patients with MC4R mutations will have decreased BDNF, the severity of which will be associated with the degree of MC4R functional loss caused by the specific mutation(s) in each individual. To test these hypotheses, we wish to conduct cross-sectional studies to evaluate serum BDNF concentrations, metabolism, body composition, and neurocognition in: subjects with PWS, subjects with MC4R mutations and control subjects matched for age, sex, race, and BMI. If alterations in BDNF are found to be associated with PWS and/or MC4R mutations, these investigations could lead to future studies of BDNF receptor agonists as mechanism-specific pharmacologic therapy for hyperphagia and obesity in PWS and MC4R mutations, or BDNF receptor antagonists for failure-to-thrive in neonatal PWS.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subject Inclusion Criteria:

1. For PWS subjects: We will enroll 75 subjects of all ages who have diagnosis of PWS confirmed by chromosome analysis (i.e. interstitial deletion of paternally-derived chromosome 15q, uniparental maternal disomy or other chromosome 15 abnormalities). Our goal is to have 25 infants, 25 non-obese, and 25 obese subjects in order to assess the different phases associated with PWS. Subjects receiving growth hormone therapy may enroll if the dose has been stable for the preceding 6 months.
2. For MC4R subjects: We will screen up to 200 subjects for mutations of MC4R and enroll 50 subjects of all ages who have diagnosis of homozygous or heterozygous MC4R mutation confirmed by sequencing of the MC4R gene. Both functional-altering (N=25) and non-pathologic (N=25) mutations will be included.
3. For control subjects: We will enroll 125 subjects of all ages who match with PWS or MC4R subjects by age (plus-minus 10%), sex, race, and BMI percentile (plus-minus10%).

EXCLUSION CRITERIA:

Subject Exclusion Criteria:

1. For all subjects:

   1. Pregnancy
   2. Individuals who have, or whose parent or guardians have, current substance abuse or a psychiatric disorder or other condition which, in the opinion of the investigators, would impede competence or compliance or possibly hinder completion of the study
   3. If age >12 months, greater than 2% body weight loss in preceding 6 months
   4. Anorexiant or weight loss medication use in preceding 6 months
2. For control subjects:

   1. Chronic medical conditions anticipated to affect results or impede study participation
   2. Medication use will be reviewed on a case-by-case basis by the Principal Investigator to determine eligibility

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-01-09; Study Completion 2014-12-12

PRIMARY OUTCOMES:
Serum brain-derived neurotrophic factor concentration

SECONDARY OUTCOMES:
Body Composition, Cognitive Function

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (2):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- University of Alberta, Alberta, Canada

REFERENCES:
- [Background] Cohen-Cory S, Kidane AH, Shirkey NJ, Marshak S. Brain-derived neurotrophic factor and the development of structural neuronal connectivity. Dev Neurobiol. 2010 Apr;70(5):271-88. doi: 10.1002/dneu.20774. PMID 20186709
- [Background] Wisse BE, Schwartz MW. The skinny on neurotrophins. Nat Neurosci. 2003 Jul;6(7):655-6. doi: 10.1038/nn0703-655. No abstract available. PMID 12830151
- [Background] Xu B, Goulding EH, Zang K, Cepoi D, Cone RD, Jones KR, Tecott LH, Reichardt LF. Brain-derived neurotrophic factor regulates energy balance downstream of melanocortin-4 receptor. Nat Neurosci. 2003 Jul;6(7):736-42. doi: 10.1038/nn1073. PMID 12796784
- [Derived] Han JC, Reyes-Capo DP, Liu CY, Reynolds JC, Turkbey E, Turkbey IB, Bryant J, Marshall JD, Naggert JK, Gahl WA, Yanovski JA, Gunay-Aygun M. Comprehensive Endocrine-Metabolic Evaluation of Patients With Alstrom Syndrome Compared With BMI-Matched Controls. J Clin Endocrinol Metab. 2018 Jul 1;103(7):2707-2719. doi: 10.1210/jc.2018-00496. PMID 29718281